CLINICAL TRIAL: NCT02812836
Title: 3D High Resolution Manometry and Balloon Expulsion Test in Diagnosis of Dyssynergic Defecation in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Marcin Banasiuk, PhD, Medical University of Warsaw
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Banasiuk 2016B
Record Dates: First submitted 2016-06-22; First posted 2016-06-24 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Children; Constipation
Keywords: anorectal manometry; children; constipation
MeSH Terms: conditions — Constipation | interventions — Manometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Manometry (Other): All patients will be investigated by anorectal manometry and after the procedure with balloon expulsion test as previously described.
  Interventions: Device: Manometry

INTERVENTIONS:
Device: Manometry — Each patient will be investigated first by anorectal manometry, standard protocol of conventional parameters will be recorded such as: resting pressure, squeeze pressure, bear down manoeuver, thresholds of sensation and threshold of recto anal inhibitory reflex. 3D picture of anal canal will be recorded. After that balloon with 50 ml of water will be inserted into the rectum and patient will be asked to expel the device within 1 min in privacy.
  Other Names: Balloon

SUMMARY:
Anorectal 3D manometry (3D HRAM) is the most advanced version of manometric equipment that measures pressures along the anal canal in a very detailed manner. It provides complete data about pressure profile of anorectum and may indicate impaired defecation dynamics. Balloon expulsion test (BET) is a cheap, easy way to diagnose constipation as the result of outlet obstruction.

Our aim is to compare this two methods of diagnosis of dyssynergic defecation and to find the correlation between this diagnostic equipment.

DETAILED DESCRIPTION:
Patients with the diagnosis of constipation will be enrolled in the study. Each patient will be investigated by anorectal manometry and after the procedure BET will be performed at the same day.

During anorectal manometry conventional manometric parameters will be recorded, such as resting pressure, squeeze pressure, bear down manoeuver, thresholds of sensation and threshold of recto anal inhibitory reflex. 3D picture of anal canal will be recorded.

After the manometry standard BET will be performed. The balloon will be inserted into the rectum and patient will be asked to expel it in private during 1 min.

Data from manometry will be correlated with the success rate of BET.

ELIGIBILITY:
Inclusion Criteria:

* Constipation
* Parental agreement

Exclusion Criteria:

* after surgery on lower gastrointestinal tract
* diagnosis of inflammatory bowel disease
* diagnosis of other disorder that may affect anorectum function
* parental disagreement

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between percent of dyssynergic defecation diagnosed by the manometry and BET. | 30 min
  Percent of patients with the diagnosis of dyssynergic defecation made by BET and according to manometric equipment.

SECONDARY OUTCOMES:
Bear down manoeuver pressure differential | 1 min
  Pressures of rectum and anal canal during bear down manoeuver will be recorded 3 times. Patients will be classified as dyssynergic defecation type. Correlation between the type and the result of BET will be evaluated.
puborectalis muscle pressure | 1 min
  3D picture of anal canal will be recorded and pressure of puborectalis muscle will be recorded during rest and squeeze. The level of pressure will be correlated with the result of BET

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Banasiuk, PhD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of Pediatric Gastroenterology and Nutrition, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No